CLINICAL TRIAL: NCT03678649
Title: A Prospective Randomized Controlled Clinical Trial of Capecitabine Treatment in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck After Radiotherapy: Phase II Study
Brief Title: A Prospective Randomized Trial of Capecitabine Treatment in Patients With HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2018-HNC01
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms;Capecitabine
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment arm (Experimental): 1000-1250 mg/m2 orally twice daily for 14 days followed by a 1-week rest period, given as 3- week cycles for a total of 6 cycles .
  it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Capecitabine
- the control arm (No Intervention): clinical observation

INTERVENTIONS:
Drug: Capecitabine — 1000-1250 mg/m2 orally twice daily for 14 days followed by a 1-week rest period, given as 3- week cycles for a total of 6 cycles .
  Arms: the treatment arm

SUMMARY:
This prospective randomized controlled clinical Trial will be performed in patients with locally advanced squamous cell carcinoma of the head and neck. The objectives of the trial are to compare the efficacy and safety of Capecitabine treatment with placebo as adjuvant therapy to patients who have received radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. histologically type： squamous cell carcinoma
2. head and neck squamous cell carcinoma (HNSCC), Tumor staged as III to IVb (according to the 8th AJCC edition).
3. Eastern cooperative oncology group (ECOG) performance status 0 or 1
4. Age between 18 and 65 years old
5. Prior treatment with chemo-radiotherapy (CRT) based Platinum drugs.
6. Adequate marrow: WBC count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
7. Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ 1.5ULN.
8. Adequate renal function: creatinine clearance ≥60 ml/min.
9. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Nasopharyngeal carcinoma and/or salivary gland carcinoma.
2. Any other malignancy (except for primaries, appropriately treated superficial basal cell skin cancer and surgically cured cervical cancer in situ)
3. currently recurrent of metastatic disease
4. received research drug in 4 weeks
5. Prior treatment with epidermal growth factor receptor (EGFR)-targeted small molecules, EGFR-targeted antibodies, and/or any investigational agents for HNSCC
6. Severe hematological abnormality and intolerance to chemotherapy
7. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.
8. Pregnancy or breast feeding
9. patients who cannot obey to completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS (progression free survival) | 3-year
  PFS is calculated from the date of randomisation to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from the date of randomization to death from any cause.
Locoregional failure-free survival | 3-year
  Locoregional failure-free survival is calculated from the date of randomization to the first locoregional failure.
Distant failure-free survival | 3-year
  Distant failure-free survival is calculated from the date of randomization to the first remote failure.
QoL(quality of life) | 3-year
  Changes in quality of life were assessed by EORTC C30; QLQ-H&N35 (V1.0)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No